CLINICAL TRIAL: NCT04386057
Title: Phase II Trial of ERK Inhibition Alone and in Combination With Autophagy Inhibition in Patients With Metastatic Pancreatic Cancer
Brief Title: LY3214996 +/- HCQ in Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kimberly Perez, MD (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Kimberly Perez, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-529
Record Dates: First submitted 2020-05-10; First posted 2020-05-13 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer; Advanced Cancer
Keywords: Pancreatic Cancer; Advanced Cancer; Extracellular Signal-Regulated Kinases; Cell Growth Inhibitors
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Hydroxychloroquine; LY3214996

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Lead-In Cohort (Experimental): The research study procedures include screening for eligibility and study treatment. Study treatment will include evaluations, biopsies, and follow up visits. A treatment cycle will be defined as 28 consecutive days. Treatment will be administered on an outpatient basis.
  Test the safety of study drugs in combination and define dose levels.
  * LY3214996
  * HCQ
  Interventions: Drug: Hydroxychloroquine Sulfate; Drug: LY3214996
- LY3214996 and HCQ Combination (Experimental): The research study procedures include screening for eligibility and study treatment. Study treatment will include evaluations, biopsies, and follow up visits. A treatment cycle will be defined as 28 consecutive days. Treatment will be administered on an outpatient basis. Combined dosage per determined Lead-In Cohort
  * LY3214996
  * HCQ
  Interventions: Drug: Hydroxychloroquine Sulfate; Drug: LY3214996
- LY3214996-Monotherapy (Experimental): The research study procedures include screening for eligibility and study treatment. Study treatment will include evaluations, biopsies, and follow up visits. A treatment cycle will be defined as 28 consecutive days.Treatment will be administered on an outpatient basis.
  -LY3214996
  Interventions: Drug: LY3214996
- Cross Over Arm (Experimental): Participants who are enrolled to Arm 2 who experience radiologic disease progression on monotherapy will have the option to cross-over to receive treatment with the combination. Crossover will occur at the treating investigator's discretion following consultation and approval from the overall principal investigator. Combined dosage per determined Lead-In Cohort
  * LY3214996
  * HCQ
  Interventions: Drug: Hydroxychloroquine Sulfate; Drug: LY3214996

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — HCQ will be administered by mouth twice daily continuously throughout each treatment per 28 day cycle
  Other Names: Plaquenil®); HCQ
  Arms: Cross Over Arm; LY3214996 and HCQ Combination; Safety Lead-In Cohort
Drug: LY3214996 — LY3214996-daily oral dosage per protocol per 28 day cycle

SUMMARY:
This study is evaluating the safety and efficacy of combining the study drug LY3214996 with hydroxychloroquine sulfate (HCQ) in patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
* This is an open label, randomized, two arm, phase II with safety lead- in study exploring the anti-tumor activity of the extracellular signal-regulated kinase (ERK) inhibitor LY3214996 with and without hydroxychloroquine (HCQ) in patients with advanced pancreatic cancer.
* The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

  * The safety lead-in will test the safety of a combination of investigational drugs and also try to define appropriate dosage. The names of the study drugs involved in this study are:

    * LY3214996
    * Hydroxychloroquine Sulfate (HCQ)
  * Following completion of a brief combination treatment safety lead-in cohort, participants will be randomized 1:1 for enrollment to one of two treatment arms:

    * Arm 1: receiving combination treatment with LY3214996 and HCQ
    * Arm 2: receiving monotherapy treatment with LY3214996

It is expected that about 52 people will take part in this research study

The U.S. Food and Drug Administration (FDA) has not approved LY3214996 as a treatment for any disease.

The U.S. Food and Drug Administration (FDA) has not approved HCQ for your specific disease but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed adenocarcinoma or poorly differentiated carcinoma of the pancreas.
* Age ≥ 18 years.
* ECOG performance status ≤ 1
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for nonnodal lesions and short axis for nodal lesions) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan, MRI, or calipers by clinical exam.
* Participants must have received at least one but no more than two prior lines of systemic therapy for metastatic pancreatic cancer. Perioperative treatment (chemotherapy and/or radiation) is not considered a prior line of therapy.
* Participants must have adequate organ and marrow function as defined below:

  * Absolute Neutrophil Count ≥ 1,500/mcL
  * Platelet Count ≥ 100,000/mcL
  * Total Bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  * AST (SGOT) / ALT(SGPT) ≤ 2.5 × institutional ULN, OR
  * AST (SGOT) / ALT (SGPT) ≤ 5 × institutional ULN if elevation is a result of metastases
  * Creatinine ≤ 1.5 × institutional ULN, OR
  * Creatinine Clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above 1.5 × institutional normal (calculated via the Cockcroft-Gault equation)
* The effects of LY3214996 or HCQ on the developing human fetus are unknown. For this reason and because anti-cancer agents are known to be teratogenic, women of child bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of LY3214996 or HCQ administration.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow and retain oral medication
* Baseline QTcB of ≤ 470 msec on screening EKG.
* Participants must be able and willing to undergo the pre-treatment biopsy procedure, and have a cancer site amenable to biopsy.

Exclusion Criteria:

* Participants with pancreatic histologies other than adenocarcinoma or poorly differentiated carcinoma, such as neuroendocrine or acinar cell carcinoma.
* Participants who have received a prior MAPK pathway inhibitor, including but not limited to LY3214996.
* Participants who have had systemic chemotherapy, other investigational therapy, or immunotherapy within 3 weeks prior to the first dose of study medication.
* Participants who have received oral tyrosine kinase inhibitors (TKIs) within 5 half-lives of the first dose of study medication.
* Participants who have received radiation therapy within 2 weeks prior to the first dose of study medication.
* Participants who have had major surgery within 4 weeks prior to the first dose of study medication.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to LY3214996 or HCQ. Individuals with a history of a different malignancy are ineligible with the following exceptions: individuals who have been treated and are disease-free for a minimum of 3 years prior to study enrollment, or individuals who are deemed by the treating investigator to be at low risk for disease recurrence. Additionally, individuals with the following cancers are eligible if diagnosed and curatively treated within the past 3 years: basal or squamous cell carcinomas of the skin, and breast or cervical carcinomas in situ.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because LY3214996 and HCQ are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LY3214996 or HCQ, breastfeeding should be discontinued if the mother is treated with LY3214996 or HCQ. A negative serum pregnancy test is required for women of childbearing potential prior to the first dose of study medication.
* Participants who are known to be seropositive for human immunodeficiency virus (HIV) or hepatitis B or C.
* Participants with a history or findings of central or branch retinal artery or venous occlusion with significant vision loss, or other retinal diseases causing visual impairment or would likely cause visual impairment over the time period of the study, as assessed by an ophthalmologist.
* Participants with a known personal or family history of long QT syndrome.
* Participants with known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Participants who are known at the time of trial enrollment to require concomitant treatment with strong CYP3A4 inhibitors or inducers. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2024-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Perez, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Lead-In Cohort: Dose Level 0 (400mg LY3214996): The research study procedures include screening for eligibility and study treatment. Study treatment will include evaluations, biopsies, and follow up visits. A treatment cycle will be defined as 28 consecutive days. Treatment will be administered on an outpatient basis.
  Test the safety of study drugs in combination and define dose levels.
  * LY3214996
  * HCQ
  Hydroxychloroquine Sulfate: HCQ will be administered by mouth twice daily continuously throughout each treatment per 28 day cycle. All dose levels will have a 400mg HCQ dose.
  LY3214996: LY3214996-daily oral dosage per protocol per 28 day cycle. Dose level 0 will have a 400mg LY3214996 dose.
- Safety Lead-In Cohort: Dose Level -1 (200mg LY3214996): The research study procedures include screening for eligibility and study treatment. Study treatment will include evaluations, biopsies, and follow up visits. A treatment cycle will be defined as 28 consecutive days. Treatment will be administered on an outpatient basis.
  Test the safety of study drugs in combination and define dose levels.
  * LY3214996
  * HCQ
  Hydroxychloroquine Sulfate: HCQ will be administered by mouth twice daily continuously throughout each treatment per 28 day cycle. All dose levels will have a 400mg HCQ dose.
  LY3214996: LY3214996-daily oral dosage per protocol per 28 day cycle. Dose level -1 will have a 200mg LY3214996 dose.
- LY3214996 and HCQ Combination: The research study procedures include screening for eligibility and study treatment. Study treatment will include evaluations, biopsies, and follow up visits. A treatment cycle will be defined as 28 consecutive days. Treatment will be administered on an outpatient basis. Combined dosage per determined Lead-In Cohort
  * LY3214996
  * HCQ
  Hydroxychloroquine Sulfate: HCQ will be administered by mouth twice daily continuously throughout each treatment per 28 day cycle
  LY3214996: LY3214996-daily oral dosage per protocol per 28 day cycle
- LY3214996-Monotherapy: The research study procedures include screening for eligibility and study treatment. Study treatment will include evaluations, biopsies, and follow up visits. A treatment cycle will be defined as 28 consecutive days.Treatment will be administered on an outpatient basis.
  -LY3214996
  LY3214996: LY3214996-daily oral dosage per protocol per 28 day cycle
- Cross Over Arm: Participants who are enrolled to Arm 2 who experience radiologic disease progression on monotherapy will have the option to cross-over to receive treatment with the combination. Crossover will occur at the treating investigator's discretion following consultation and approval from the overall principal investigator. Combined dosage per determined Lead-In Cohort
  * LY3214996
  * HCQ
  Hydroxychloroquine Sulfate: HCQ will be administered by mouth twice daily continuously throughout each treatment per 28 day cycle
  LY3214996: LY3214996-daily oral dosage per protocol per 28 day cycle
Period: Overall Study
Arm/Group | Safety Lead-In Cohort: Dose Level 0 (400mg LY3214996) | Safety Lead-In Cohort: Dose Level -1 (200mg LY3214996) | LY3214996 and HCQ Combination | LY3214996-Monotherapy | Cross Over Arm
Started | 7 | 6 | 20 | 16 | 3
Completed | 7 | 6 | 20 | 16 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were collected for all participants enrolled on the study (52). Characteristics are separated by Arm (7 in safety lead-in dose level 0, 6 in safety lead-in dose level -1, 20 in combination therapy, 16 in monotherapy, and 3 in crossover).
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Lead-In Cohort: Dose Level 0 (400mg LY3214996) | Safety Lead-In Cohort: Dose Level -1 (200mg LY3214996) | LY3214996 and HCQ Combination | LY3214996-Monotherapy | Cross Over Arm | Total
Number analyzed (Participants) | 7 | 6 | 20 | 16 | 3 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 10 | 3 | 0 | 16
  >=65 years | 6 | 4 | 10 | 13 | 3 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 7 | 6 | 1 | 19
  Male | 3 | 5 | 13 | 10 | 2 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 6 | 6 | 17 | 16 | 2 | 47
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 0 | 0 | 4
  White | 4 | 5 | 17 | 14 | 3 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 20 | 16 | 3 | 52

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: Anti-tumor activity will be measured via disease control rate (DCR), which will be defined as the proportion of patients with complete response (CR), partial response (PR) or stable disease (SD) that persists for ≥ 4 months. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameters of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 28 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Lead-In Cohort: Dose Level 0 (400mg LY3214996) | Safety Lead-In Cohort: Dose Level -1 (200mg LY3214996) | LY3214996 and HCQ Combination | LY3214996-Monotherapy | Cross Over Arm
Number analyzed (Participants) | 7 | 6 | 20 | 16 | 3
Participants | 0 | 1 | 1 | 1 | 0

2. Primary Outcome: Dose Limiting Toxicity-Lead In
Description: Dose Limiting Toxicity-Lead In
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Lead-In Cohort: Dose Level 0 (400mg LY3214996) | Safety Lead-In Cohort: Dose Level -1 (200mg LY3214996)
Number analyzed (Participants) | 7 | 6
Participants | 2 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the number of participants who had a complete or partial response at any time during treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameters of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 28 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Lead-In Cohort: Dose Level 0 (400mg LY3214996) | Safety Lead-In Cohort: Dose Level -1 (200mg LY3214996) | LY3214996 and HCQ Combination | LY3214996-Monotherapy | Cross Over Arm
Number analyzed (Participants) | 7 | 6 | 20 | 16 | 3
Participants | 0 | 0 | 1 | 0 | 0

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study . The sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesion and/or unequivocal progression of existing non-target lesions are also considered progression. Unequivocal progression should not normally trump target lesion status and must be representative of overall disease status change, not a single lesion increase.
Time Frame: time from randomization (or registration) to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation up to 28 Months
Population: PFS (months) was calculated for participants only in the randomized arms (including crossovers in their original arm) as an Intention to Treat Analysis (ITT). Analyses were not completed for participants in the safety lead-in cohort, as this cohort was intended to evaluate safety only; not efficacy. Only 14 participants were evaluable for PFS in Arm A and 17 were evaluable in Arm B. These numbers differ slightly to the overall number of participants due to missing data and adding crossovers.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LY3214996 and HCQ Combination | LY3214996-Monotherapy
Number analyzed (Participants) | 14 | 17
months | 1.3 [0.8 to 1.8] | 1.9 [1.6 to 2.4]

5. Secondary Outcome: Overall Survival (OS)
Description: Kaplan and Meier to assess Overall survival (OS)
Time Frame: Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive. OS was calculated for a median of 115 days, ranging from 18 - 327 days.
Population: OS (months) was calculated for participants only in the randomized arms (including crossovers in their original arm) as an Intention to Treat Analysis (ITT). Analyses were not completed for participants in the safety lead-in cohort, as this cohort was intended to evaluate safety only; not efficacy. Only 17 participants were evaluable from Arm A and 19 were evaluable from Arm B. These numbers differ slightly to the overall number of participants due to missing data and adding crossovers.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LY3214996 and HCQ Combination | LY3214996-Monotherapy
Number analyzed (Participants) | 17 | 19
months | 2.4 [1.3 to 5.8] | 4.7 [3.1 to 5.7]

ADVERSE EVENTS:
Time Frame: Adverse Events were reviewed between the initial dose of study treatment (first patient treated June 2020) and 30 days of the last dose of treatment (last patient September 2023). Participants were assessed for AEs for a median of 67 days (range 31-141 days). All-cause mortality was assessed from date of randomization to death of any cause or last known date alive, for a median of 115 days (range 18-327 days).
Description: After completion of the 30 day follow up period, participants will continue to be followed for 6 months after removal of protocol therapy or until death for survival status only. Considering this, the total length of study differs from the total adverse event collection time frame.
Arm/Group | Safety Lead-In Cohort: Dose Level 0 (400mg LY3214996) | Safety Lead-In Cohort: Dose Level -1 (200mg LY3214996) | LY3214996 and HCQ Combination | LY3214996-Monotherapy | Cross Over Arm
All-Cause Mortality (participants affected / at risk) | 7/7 | 6/6 | 18/20 | 13/16 | 3/3
Serious Adverse Events (participants affected / at risk) | 7/7 | 3/6 | 6/20 | 4/16 | 1/3
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 16/20 | 16/16 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Lead-In Cohort: Dose Level 0 (400mg LY3214996) (N=7) | Safety Lead-In Cohort: Dose Level -1 (200mg LY3214996) (N=6) | LY3214996 and HCQ Combination (N=20) | LY3214996-Monotherapy (N=16) | Cross Over Arm (N=3)
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
CPK increased (Investigations) | 0 | 0 | 1 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0
Fever (General disorders) | 1 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Lead-In Cohort: Dose Level 0 (400mg LY3214996) (N=7) | Safety Lead-In Cohort: Dose Level -1 (200mg LY3214996) (N=6) | LY3214996 and HCQ Combination (N=20) | LY3214996-Monotherapy (N=16) | Cross Over Arm (N=3)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 7 | 6 | 3
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 7 | 9 | 2
Alkaline phosphatase increased (Investigations) | 2 | 2 | 8 | 4 | 2
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 9 | 8 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 4 | 7 | 5 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 6 | 8 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2 | 0
Belching (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 3 | 5 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blurred vision (Eye disorders) | 0 | 0 | 0 | 1 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac troponin T increased (Investigations) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 3 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 4 | 4 | 9 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0
CPK increased (Investigations) | 4 | 1 | 4 | 1 | 1
Creatinine increased (Investigations) | 1 | 1 | 3 | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 4 | 3 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 4 | 7 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Edema limbs (General disorders) | 1 | 1 | 2 | 1 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 5 | 0 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Facial muscle weakness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 2 | 0
Fatigue (General disorders) | 2 | 5 | 11 | 10 | 2
Fever (General disorders) | 0 | 0 | 3 | 4 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Generalized edema (General disorders) | 0 | 0 | 1 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 5 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 3 | 7 | 6 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 5 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 4 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 9 | 6 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 2 | 1
Investigations - Other, specify (Investigations) | 0 | 0 | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 2 | 6 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 3 | 12 | 12 | 3
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Night sweats (General disorders) | 0 | 0 | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 1 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Periorbital edema (Eye disorders) | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 0 | 2 | 0
Platelet count decreased (Investigations) | 4 | 1 | 4 | 10 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 4 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Thrush (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 3 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 7 | 8 | 1
Weight gain (Investigations) | 1 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 1 | 2 | 2 | 1
White blood cell decreased (Investigations) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT04386057/Prot_SAP_000.pdf